CLINICAL TRIAL: NCT07360132
Title: A Randomized, Double-Blind, Multicenter Phase III Clinical Study of HB0025 Combined With Chemotherapy Versus Pembrolizumab Combined With Chemotherapy for the First-Line Treatment of Advanced or Metastatic Squamous Non-Small Cell Lung Cancer
Brief Title: Phase III Clinical Study of HB0025 Combined With Chemotherapy Versus Pembrolizumab Combined With Chemotherapy for the First-Line Treatment of Advanced Squamous Non-Small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Huaota Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HB0025-C-0302
Record Dates: First submitted 2026-01-13; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Squamous Non-small Cell Lung Cancer
Keywords: HB0025; sq-NSCLC; Fiest Line treatment
MeSH Terms: interventions — Carboplatin; Paclitaxel

STUDY DESIGN:
Intervention Model Description: It is planned to enroll approximately 480 subjects, and they will be randomly divided into groups at a ratio of 1:1. The treatment is administered once every 3 weeks (Q3W). After 4 cycles of treatment, patients will proceed to receive maintenance therapy with HB0025 or pembrolizumab alone (also Q3W).
  Experimental group: HB0025 combined with chemotherapy Paclitaxel plus Platinum; Control group: pembrolizumab combined with chemotherapy Paclitaxel plus Platinum.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HB0025 (Experimental): HB0025 combined with Carboplatin Injection plus Paclitaxel Injection, IV, every 3 weeks(Q3W)
  Interventions: Drug: Carboplatin Injection; Drug: Paclitaxel Injection
- Pembrolizumab (Active Comparator): pembrolizumab combined with Carboplatin Injection plus Paclitaxel Injection, IV every 3 weeks (Q3w)
  Interventions: Drug: Carboplatin Injection; Drug: Paclitaxel Injection

INTERVENTIONS:
Drug: Carboplatin Injection — 10mL:100mL, Q3W
Drug: Paclitaxel Injection — 5ml:30mg, Q3W

SUMMARY:
This study is a randomized, controlled, double-blind, multi-center phase III registration clinical trial, aiming to observe, compare and evaluate the efficacy and safety of HB0025 combined with paclitaxel + carboplatin compared with pembrolizumab combined with paclitaxel + carboplatin as the first-line treatment for locally advanced or metastatic squamous NSCLC.

The study subjects are patients with locally advanced or metastatic squamous non-small cell lung cancer (NSCLC) who have not received systemic anti-tumor treatment before. The study will use the PFS evaluated by BICR as the primary endpoint, and plan to enroll approximately 480 subjects, with the proportion of locally advanced subjects not exceeding 10%.

The subjects were fully informed and signed the informed consent form. If they met the inclusion criteria but did not meet the exclusion criteria, they were randomly assigned in a 1:1 ratio to receive HB0025 combined with chemotherapy Paclitaxel plus Platinum (experimental group) or pembrolizumab combined with chemotherapy Paclitaxel plus Platinum (control group). Both were administered once every 3 weeks (Q3W). After 4 cycles of treatment, Enter HB0025 or pembrolizumab monotherapy maintenance treatment (Q3W) until the investigator determines that there is no longer any clinical benefit (based on the RECIST v1.1 imaging assessment and comprehensive clinical symptom assessment by the investigator), intolerable toxicity occurs, 24 months of study treatment is completed, or other treatment termination criteria in the protocol are met. Whichever occurs first shall prevail.

DETAILED DESCRIPTION:
The random stratification factors of this study are as follows:

* Disease stage: ⅢB/ⅢC stage vs Ⅳ stage;
* PD-L1 expression score indicator (tumor cell positive proportion score TPS): <1%, 1%-49%, ≥50%;
* Hepatic metastasis or brain metastasis: Yes vs No. This study uses the RECIST v1.1 standard to conduct regular tumor response assessments for the subjects. Tumor assessment are conducted at the 6th week (±7 days), the 12th week (±7 days), and every 9 weeks thereafter (±7 days) within 48 weeks after the first administration of the drug; and every 12 weeks thereafter (±7 days). If the subject stops the study treatment due to reasons other than disease progression or death, the tumor assessment should continue according to the fixed schedule until imaging progression or termination of the study (the latter occurring is the criterion), initiation of new anti-tumor treatment, loss to follow-up, death, withdrawal of informed consent, or study completion, whichever occurs first. After the first imaging progression, if the investigator believes that the subject can still benefit from continued treatment and meets the criteria listed in the protocol for continuing treatment, the subject can continue with the original treatment plan until no clinical benefit is observed (assessed by the investigator). If the subject stops the study treatment for reasons other than the above (such as occurrence of intolerable adverse events, or the subject has received 24 months of HB0025 or pembrolizumab treatment, or other reasons for stopping treatment, etc.), a tumor assessment should be conducted before terminating the study. The investigator can conduct unplanned (with an interval of at least 4 weeks greater than the previous assessment) tumor assessments in cases of suspected disease progression or other necessary circumstances. The sponsor will collect all the imaging data of the subjects for BICR assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Able to fully understand and voluntarily sign the informed consent form, and willing and able to comply with the clinical study procedures and follow-up visits.
2. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0-1.
3. Expected survival ≥ 12 weeks.
4. Histologically or cytologically confirmed locally advanced (Stage IIIB/IIIC) or metastatic (Stage IV) non-small cell lung cancer (NSCLC) (confirmed per the 9th Edition of the TNM Staging System for Lung Cancer by the Union for International Cancer Control [UICC] and the American Joint Committee on Cancer [AJCC]) that is inoperable for radical resection and ineligible for radical concurrent/sequential chemoradiotherapy or immunotherapy as consolidation treatment.

Note: For subjects with locally advanced (Stage IIIB/IIIC) NSCLC who are inoperable for radical resection and ineligible for radical concurrent/sequential chemoradiotherapy or immunotherapy as consolidation treatment, an assessment by relevant specialist physicians and provision of written documentation are required for confirmation.

6. No previous systemic anti-tumor treatment for locally advanced or metastatic squamous NSCLC [For subjects who have received adjuvant/neoadjuvant therapy for the purpose of cure for non-metastatic disease or radical concurrent/sequential chemoradiotherapy for locally advanced disease (including subjects receiving PD-1/L1 inhibitors), If disease progression occurs more than 12 months after the end of the last treatment, one is eligible to participate in this study.

7. Subjects must provide tumor tissue samples (archived or freshly obtained) collected at or after the diagnosis of locally advanced or metastatic tumor for central laboratory testing of PD-L1 expression.

Note:The following samples are not accepted: fine-needle aspiration samples (without intact tissue structure, only cell suspensions or smears), brush cytology samples, cell smears from centrifuged pleural effusion drainage, bronchoalveolar lavage fluid samples, and bone lesions without soft tissue components or decalcified bone tumor samples.

8. No sensitive EGFR mutations or ALK gene rearrangements. Prior tissue-based test reports for EGFR and ALK status must be provided. If the test reports do not meet the study requirements or are unavailable, tumor tissue samples must be provided for assessment of EGFR and ALK status (tested by a local laboratory recognized by the study site or the central laboratory) before enrollment.

Note: For subjects with squamous NSCLC (excluding mixed-type NSCLC, e.g., adenosquamous carcinoma) who have a smoking history or are current smokers, if the prior EGFR and ALK status is unknown, testing for these markers is not required before enrollment, and they will be deemed negative.

9. At least one measurable (non-brain metastatic) lesion per RECIST v1.1 criteria, which is suitable for repeated and accurate measurement. Tumor lesions previously treated with radiotherapy or other local therapies cannot be designated as target lesions, unless:

* The lesion is the only measurable lesion, and the investigator can provide imaging evidence (before and after local treatment) confirming clear disease progression of the lesion after local treatment;
* The lesion used for fresh tissue biopsy is the only measurable lesion. 10. Confirmed adequate organ function, as evidenced by meeting the following laboratory parameters: 1) Hematology (no receipt of blood component transfusion or hematopoietic growth factor support within 14 days before screening tests):

  1. Absolute Neutrophil Count (ANC) ≥ 1.5 × 10⁹/L;
  2. Platelet Count (PLT) ≥ 100 × 10⁹/L;
  3. Hemoglobin (HGB) ≥ 90 g/L; 2) Renal function:

  a) Serum Creatinine (Scr) ≤ 1.5 × Upper Limit of Normal (ULN), and Creatinine Clearance (Ccr) ≥ 50 mL/min (calculated using the Cockcroft-Gault formula); b) Urine protein < 2+; if urine protein ≥ 2+, 24-hour urine protein excretion must be < 1 g; 3) Hepatic function:
  1. Serum Total Bilirubin (TBiL) ≤ 1.5 × ULN;
  2. Serum Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) ≤ 2.5 × ULN; for subjects with liver metastasis, ALT and AST ≤ 5 × ULN;
  3. Serum Albumin (ALB) ≥ 30 g/L; 4) Coagulation function: Prothrombin Time (PT), Activated Partial Thromboplastin Time (APTT), and International Normalized Ratio (INR) ≤ 1.5 × ULN (for subjects receiving anticoagulant therapy, the investigator must confirm that INR, APTT, and PT are within the safe and effective therapeutic range); 5) Cardiac function: Left Ventricular Ejection Fraction (LVEF) ≥ 50% 11. The toxicity of previous treatment has been restored to grade 0 or 1 of NCI CTCAE version 5.0, or the level specified in the inclusion/exclusion criteria (except for alopecia). Note: For subjects who experience irreversible toxicity and whose condition is not expected to worsen after administration of the study drug (such as those with hearing loss), they may be included in the study after consultation with medical monitors.

     12. Female and male subjects of childbearing potential must agree to use effective contraceptive measures from the screening period until 90 days after the last dose of study treatment. Discussion with the investigator is required to determine whether contraception can be discontinued after this period. Female subjects must not be breastfeeding. Female subjects of childbearing potential must have a negative serum pregnancy test result within 7 days before randomization.

     Exclusion Criteria:
     1. Histologically confirmed presence of any small cell carcinoma, neuroendocrine carcinoma, or sarcoma components [mixed-type NSCLC (e.g., adenosquamous carcinoma) is permitted for enrollment].
     2. Known presence of driver gene alterations with approved first-line therapeutic options, such as sensitive EGFR mutations, ALK fusion, ROS1 fusion, BRAF V600 mutation, NTRK fusion, MET exon 14 skipping mutation, or RET fusion.
     3. History of a second primary malignancy within 3 years before Randomization (enrollment is permitted for other malignancies cured by local treatment, e.g., carcinoma in situ of the cervix, localized cutaneous squamous cell carcinoma, basal cell carcinoma, ductal carcinoma in situ of the breast, < T1 urothelial carcinoma, and papillary microcarcinoma of the thyroid).
     4. Symptomatic central nervous system (CNS) metastasis; or diameter of brain metastases ≤ 1.5 cm, or receipt of CNS radiotherapy within 2 weeks before randomization; or anticipated need for CNS radiotherapy during the first treatment cycle after randomization. Subjects with asymptomatic CNS metastasis or symptomatically stable CNS metastasis (≥ 2 weeks before randomization) are permitted for enrollment only if all the following criteria are met:

        * No increase in lesion size or new lesions after treatment; ② No history of intracranial hemorrhage;

          * Discontinuation of corticosteroid therapy > 3 days before randomization;

            * Diameter of brain metastases < 1.5 cm.
     5. Prior receipt of immunotherapy, including immune checkpoint inhibitors (e.g., anti-PD-1/L1/L2, anti-CTLA-4 agents), immune checkpoint agonists (e.g., ICOS, CD40, GITR, OX40, CD137 agents), or cellular immunotherapy, or any treatment targeting the tumor immune mechanism. Additionally, for subjects who received PD-(L)1 inhibitors in the neoadjuvant/adjuvant setting or as consolidation therapy after definitive chemoradiotherapy, enrollment may be permitted (with sponsor approval) if disease progression occurs > 12 months after the last dose of prior treatment.
     6. Prior receipt of systemic anti-angiogenic therapy, including but not limited to bevacizumab and its biosimilars, Endostar, small-molecule TKIs, and ramucirumab.
     7. Prior antineoplastic treatment or concomitant medication use (washout period calculated from the end of the last treatment):

  <!-- -->

  1. Concurrent enrollment in another clinical trial, unless it is an observational, non-interventional clinical trial or the follow-up phase of an interventional clinical trial (defined as an interval of ≥ 4 weeks between the last dose of the previous study drug and randomization in this study);
  2. Receipt of chest radiotherapy with > 30 Gy within 180 days before randomization; non-chest radiotherapy with > 30 Gy within 4 weeks before randomization; local palliative radiotherapy with ≤ 30 Gy for non-target lesions within 2 weeks before randomization;
  3. Use of Chinese herbal medicines (with antineoplastic indications) within 1 week before randomization; receipt of non-specific immunomodulatory therapy (e.g., interleukin, interferon, thymosin, tumor necrosis factor, excluding IL-11 for thrombocytopenia treatment) within 2 weeks before randomization;
  4. Need for systemic use of corticosteroids (≥ 10 mg/day prednisone or equivalent) or other immunomodulators within 2 weeks before randomization [short-term use (≤ 7 days) for prophylaxis (e.g., contrast agent allergy) or treatment of non-autoimmune diseases (e.g., delayed hypersensitivity reaction to allergens), or topical use (e.g., intraocular, intra-articular, intranasal, or inhaled administration) is permitted].
  5. Subjects who are currently using preventive or full-dose anticoagulants or antiplatelet drugs for therapeutic purposes and have not reached a stable state before randomization will not be enrolled. According to the medical standards of the enrolling institution, as long as the INR, PT and APTT of the subjects are within the therapeutic range and they have used or are currently using anticoagulants or antiplatelet drugs, they can be enrolled.

     8. Major surgery or severe trauma within 4 weeks before the first dose of study treatment; inadequate recovery from prior surgery (as judged by the investigator); anticipated need for major surgery during the study; minor local surgery (e.g., needle biopsy, endoscopy, interventional procedure/examination, excluding vascular access establishment) within 7 days before randomization; presence of incompletely healed surgical incisions or wounds.

     9. Active autoimmune disease requiring systemic treatment (e.g., treatment with immunomodulators or corticosteroids) within 2 years before randomization, except for replacement therapy (e.g., thyroid hormone, insulin, or physiological corticosteroid replacement therapy for adrenal or pituitary insufficiency).

     10. Presence of any of the following infections:

  <!-- -->

  1. Severe infection (including but not limited to comorbidities requiring hospitalization, sepsis, or severe pneumonia) within 4 weeks before the first dose of study treatment; active infection requiring systemic anti-infective treatment (with antibiotics for ≥ 7 days) within 2 weeks before randomization;
  2. Known active tuberculosis (TB) (subjects with suspected active TB must undergo clinical examination to rule out the diagnosis);
  3. Known active syphilis infection;
  4. Has a known history of HIV;
  5. Active hepatitis B or hepatitis C; asymptomatic hepatitis B virus (HBV) carriers (HBV DNA ≤ 200 IU/ml or ≤ 1000 copies/ml or below the lower limit of detection, whichever is applicable) or subjects with clinically cured hepatitis C (HCV RNA below the lower limit of detection) are permitted for enrollment.

     Note: Anti-HBV treatment is required for HBsAg-positive subjects during the study treatment period.

     11. Known hypersensitivity to protein drugs, recombinant proteins, components of HB0025, and/or components of chemotherapy drugs (pemetrexed and carboplatin/cisplatin).

     12. Uncontrolled arterial hypertension despite standard treatment (systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg).

     13. Those with a history of non-infectious pneumonia requiring systemic corticosteroid treatment in the past, or currently having interstitial lung disease, pneumoconiosis, drug/radiation-related pneumonia that requires treatment, or those with severe functional impairment indicated by pulmonary function tests.

     14. Presence of any of the following severe comorbidities:

  <!-- -->

  1. Clinically significant bleeding (including but not limited to hemoptysis [defined as coughing up or expectorating ≥ 1 teaspoon (approximately 5 ml) of fresh blood or small blood clots, or hemoptysis without sputum; subjects with blood-tinged sputum or transient hemoptysis related to diagnostic bronchoscopy or lung biopsy are permitted], gastrointestinal bleeding, nasal bleeding [subjects with bloody nasal discharge are permitted]) within 4 weeks before the first dose of study treatment; any arterial thrombosis or embolism event, or significant vascular disease (e.g., aortic aneurysm, aortic dissection) within 180 days before the first dose of study treatment; history of deep vein thrombosis within 90 days before the first dose of study treatment;
  2. Imaging findings at screening showing: Tumor invasion of large blood vessels (e.g., central pulmonary artery, central pulmonary vein, aorta, brachiocephalic artery, common carotid artery, subclavian artery, superior vena cava); tumor invasion of vital organs (e.g., heart, trachea, esophagus, main bronchus); or imaging evidence of risk for esophagotracheal fistula or esophagopleural fistula; tumor encasement of large blood vessels with vascular stenosis; or pulmonary lesions with obvious necrosis/cavitation (as judged by the investigator to pose a bleeding risk if enrolled);
  3. History of persistent bleeding disorders or coagulation disorders (past or current);
  4. Clinically significant (e.g., active) cardiovascular or cerebrovascular disease within 180 days before the first dose of study treatment, including but not limited to unstable angina requiring hospitalization, myocardial infarction, myocarditis, cardiomyopathy, New York Heart Association (NYHA) Class ≥ II congestive heart failure, poorly controlled severe arrhythmia, transient ischemic attack (TIA), cerebrovascular accident (CVA), or vascular disease (e.g., aortic aneurysm at risk of rupture); or other cardiac impairment that may affect the safety evaluation of study drugs (e.g., poorly controlled arrhythmia, myocardial ischemia); Fridericia-corrected QT interval (QTcF) > 480 ms at screening, or history of congenital long QT syndrome or family history of the syndrome;
  5. History of conditions potentially causing gastrointestinal bleeding or perforation (e.g., gastrointestinal obstruction, acute Crohn's disease, ulcerative colitis, esophagogastric varices, gastrointestinal perforation, unhealed wound, intra-abdominal abscess, or acute gastrointestinal bleeding) within 180 days before the first dose of study treatment; subjects with chronic Crohn's disease or ulcerative colitis (excluding those who have undergone total colectomy and proctectomy) are excluded, even if in remission;
  6. History of gastrointestinal fistula or genitourinary fistula (past or current) that remains unhealed after surgical treatment;
  7. Hydronephrosis unrelieved by nephrostomy or ureteral stenting, or infected hydronephrosis/hydroureter;
  8. Current presence of third-space fluid collections (e.g., pleural effusion, pericardial effusion, abdominal/pelvic effusion) requiring repeated puncture/drainage for local management; or receipt of local drainage within 2 weeks before the first dose of study treatment;
  9. Acute exacerbation of chronic obstructive pulmonary disease within 30 days before the first dose of study treatment;
  10. Current presence of uncontrolled comorbidities, including but not limited to decompensated liver cirrhosis, nephrotic syndrome, uncontrolled metabolic disorders, severe active peptic ulcer disease or gastritis (enrollment decision requires joint discussion between the investigator and the sponsor).

      15. Pregnant or lactating women, or those planning to breastfeed during the study period.

      16. There is a known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.

      17. Live virus vaccine or attenuated live vaccine was received within 30 days before randomization, or vaccination was planned during the study period (Note: Inactivated vaccine is allowed).

      18. It is known that there is a history of mental illness, alcoholism, drug abuse or substance abuse.

      19. There have been or are currently uncontrolled metabolic disorders, local or systemic diseases not caused by tumors, secondary diseases or symptoms of tumors, abnormal laboratory tests or any treatments that may lead to higher medical risks and/or confuse research results, interfere with the subjects' participation in the entire study, or participation in the study may not be in the best interests of the subjects.

      20. Subjects who, as assessed by the researchers, are not suitable to participate in the trial for other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2028-04-10 (Estimated); Study Completion 2028-08-10 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to approximately 24 Months
  PFS is defined as the time from the date of randomization till the first documentation of disease progression (per RECIST v1.1 criteria) assessed by the investigator or death due to any cause (whichever occurs first)

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 24 Months
  OS is defined as the period from the start of randomization to the time of death due to any cause according to RECIST 1.1.
Objective Response Rate (ORR) | Up to 24 Months
  ORR is defined as the proportion of subjects achieving the best overall therapeutic effect (BOR) as complete remission (CR) or partial remission (PR) according to RECIST 1.1 by investigator.
Disease control rate (DCR) | Up to 24 Months
  DCR defined as the number of patients were confirmed CR and/or PR and/or stable disease(SD) according to RECIST 1.1 by investigator divided by the patients with at least one tumour evaluation
Duration of response (DOR) | Up to 24 Months
  DOR is defined as the time from the first record of CR or PR to the first record of disease. DOR as evaluated by investigators according to RECIST v1.1.
Time to Progression(TTP) | Up to 24 Months
  TTP is defined as the time from the time of randomization to the occurrence of disease progression according to recist 1.1 by investigator.
Objective Response Rate (ORR)-BICR | Up to 24 Months
  ORR is defined as the proportion of subjects achieving the best overall therapeutic effect (BOR) as complete remission (CR) or partial remission (PR) according to RECIST 1.1 by BICR
Disease control rate (DCR)-BICR | Up to 24 Months
  DCR defined as the number of patients were confirmed CR and/or PR and/or stable disease(SD) according to RECIST 1.1 by BICR divided by the patients with at least one tumour evaluation
Duration of response (DOR)-BICR | Up to 24 Months
  DOR is defined as the time from the first record of CR or PR to the first record of disease. DOR as evaluated by BICR according to RECIST v1.1
Time to Progression(TTP)-BICR | Up to 24 Months
  TTP is defined as the time from the time of randomization to the occurrence of disease progression according to recist 1.1 by BICR
Safety Assement | Up to 24 Months
  The incidence, severity and outcome of adverse events (AE), serious adverse events (SAE), immune-related adverse events (irAE) and adverse events of special concern (AESI) per NCI-CTCAE V5.0
Maximum serum concentration(Cmax) | Up to 24 Months
  Cmax refers to The maximum blood concentration of HB0025 after administration. - Sample concentration analysis method adopts ELISA. parameters will be calculated by Phoenix WinNonlin version 8.3.
Anti-drug antibodies (ADA) | Up to 24 Moths
  Incidence of positive anti-drug antibodies(ADA).

OTHER OUTCOMES:
PD-L1 expression | Approximately 16 months.
  Exploring the correlation between the levels of biomarkers (PD-L1) and the efficacy of combined treatment by Immunohistochemistry.

CONTACTS AND LOCATIONS:
Locations (1):
- The East Hospital Affiliated to Tongji University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided